CLINICAL TRIAL: NCT05166642
Title: Prospective, Randomized Clinical Trial Assessing Post-operative Wound Healing Complications Following Total Joint Arthroplasty When Using Bandgrip Incision Closure Compared to Standard Suture Closure
Brief Title: Bandgrip vs Traditional Sutures TJA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporary hold on recruitment
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bandgrip001
Record Dates: First submitted 2021-12-07; First posted 2021-12-22 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Sutures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bandgrip Micro-Anchor Skin Closure (Active Comparator)
  Interventions: Device: Bandgrip Micro-Anchor Wound Closure
- Standard of Care wound closure (Active Comparator): Standard Monocryl suture closure
  Interventions: Device: Suture closure

INTERVENTIONS:
Device: Bandgrip Micro-Anchor Wound Closure — This treatment group will utilize a suture closure technique for the deep dermal layers with Bandgrip being applied to the most superficial layer of the surgical incision
  Arms: Bandgrip Micro-Anchor Skin Closure
Device: Suture closure — This treatment gourd will utilize suture closure technique for all layers of the surgical incision.
  Arms: Standard of Care wound closure

SUMMARY:
Total Joint Arthroplasty (TJA) has become one of the most performed elective procedures. While the results of this procedure are often consistent with high patient satisfaction and return-to-function, wound-related complications can contribute to high-cost "bundle busters". Following surgery, wound drainage or other wound complications can lead to increased cost and decreased patient satisfaction. Secure wound closure is an important step in preventing wound-related complications. The surgical incision should be closed in a manner that prevents the wound edges from separating which could lead to possible drainage and bacterial contamination of the incision.

Traditional incision closure following TJA includes sutures. These sutures are then removed in the office. BandGrip is a wound closure device that can be used to approximate skin edges of wounds from surgical incisions and traumatic lacerations. It is a bandage-type patch with several small skin anchors that are used to hold the skin edges together. The clear microanchors are 0.029 inches in height and do not puncture through the dermis. There is no need for medical removal as the patient can remove the bandage.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female greater than 18 years of age
2. Scheduled to undergo primary total knee or total hip replacement
3. Able to read and comprehend informed consent form and comply with the follow-up evaluation schedule

Exclusion Criteria:

1. Prior surgical incision or scar in close proximity of the proposed incision (<2 cm).
2. Local skin conditions such as dermatitis, eczema, or psoriasis.
3. Active or previous infection in the skin or the hip or knee to be operated.
4. Inflammatory arthritis; connective tissue or vascular disorders or diseases that would adversely affect wound healing including the use of oral or topical corticosteroid use
5. Subject has a recent history of bleeding, coagulation and/or clotting disorders
6. Subject has a known allergy to BandGrip material (polycarbonate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with wound healing complications | From time of surgery to 30 days post-op
  All wound-related complication following surgery

SECONDARY OUTCOMES:
Closure time of surgical wound | Procedure (The time from the first skin pass with the suture needle until the time the last suture knot is tied will be recorded in seconds)
  Time (in seconds) that it takes to close the incisional wound during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedics, Philadelphia, Pennsylvania, United States